CLINICAL TRIAL: NCT00782951
Title: A Randomized, Double-blind, Active and Placebo Controlled Trial to Compare the Relative Analgesic Efficacy and Safety of a Single Intravenous Dose of ORG 28611 3 mcg/kg, Morphine Sulfate 0.12 mg/kg, and Placebo in Patients Experiencing Moderate to Severe Pain After Dental Impaction Surgery.
Brief Title: A Comparison of Analgesic Efficacy Between a Single Dose of ORG 28611, Morphine, and Placebo After Dental Impaction Surgery (Study P05800)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05800; Study 231006;; EudraCT Number: 2006-002571-40
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Org 28611 (Experimental)
  Interventions: Drug: Org 28611
- morphine sulfate (Active Comparator)
  Interventions: Drug: morphine sulfate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Org 28611 — single IV dose of Org 28611 3 mcg/kg after dental impaction surgery
  Other Names: SCH 900111
  Arms: Org 28611
Drug: morphine sulfate — single IV dose of morphine sulfate 0.12 mg/kg after dental impaction surgery
  Arms: morphine sulfate
Drug: Placebo — single IV dose of placebo after dental impaction surgery
  Arms: Placebo

SUMMARY:
Patients will receive a single intravenous (IV) infusion administered over 3 minutes of either ORG 28611 (SCH 900111), 0.12 mg/kg morphine sulphate, or placebo, within 6 hours after dental surgery, when they experience moderate to severe dental pain. Patient will then be evaluated with pain assessments at Baseline, 5, 10, 15, 30, 45, 60, and 90 minutes; and 2 through 8 hours or before rescue medication is needed.

ELIGIBILITY:
Inclusion Criteria:

* Has at least one mandibular partial or full bony impacted third molar requiring extraction. An ipsilateral maxillary third molar may also be extracted as may any adjacent supernumerary tooth (teeth)
* Is willing and able to understand and complete the pain evaluations
* Is male aged 18 to 40 years (inclusive)
* A subject, who has sexual partners of child-bearing potential, has agreed to use barrier contraception in addition to having their partner use another method for three months from the time of dosing. Also has agreed to abstain from sexual intercourse with pregnant or lactating women or to use condoms.
* Has a body mass index (BMI) less than or equal to 32 kg/m^2 and has a body weight of at least 65 kg
* Is in generally good health
* Is able to speak, read, and understand English and provide meaningful written informed consent
* Is able to remain at the research center for the entire 24-hours trial period
* Has an initial pain intensity score of at least 45-mm on a 100-mm VAS and moderate or severe pain on a 4-point categorical scale within 6 hours of the end of surgery (VAS as the primary parameter and the categorical as a secondary parameter)
* Is willing to return to the research center for the post-treatment visit 5 to 9 days after surgery and complete a day 30 SAE telephone call.

Exclusion Criteria:

* Has uncontrolled or clinically significant cardiovascular, respiratory, gastrointestinal, renal, hepatic, metabolic, hematological, or immunological disease
* Has a history of seizures, a family history of seizure disorder, or psychotic illness
* Has a known allergy or significant adverse reaction to opioids or opioid antagonists, paracetamol or ibuprofen
* Has a history of chronic opioid or cannabis use or abuse within 6 months prior to the start of this trial
* Has a positive urine drug test at screening or prior to surgery
* Has participated in a trial of an investigational drug or device within 30 days prior to the trial
* Has taken any of the following drugs within 4 hours or 5 elimination half-lives (whichever is greater) prior to dosing: aspirin, acetaminophen (paracetamol), nonsteroidal anti-inflammatory drugs (NSAIDs, COX-2 inhibitors), opioids, opioid combination drugs, sedative-hypnotics, muscle relaxants, and/or sedating antihistamines
* Has taken a long-acting analgesic (e.g., naproxen or celecoxib) or central nervous system (CNS) depressant within 12 hours prior to dosing
* Has taken a monoamine oxidase (MAO) inhibitor or tricyclic antidepressant drug within 4 weeks prior to administration of trial medication
* Has taken a selective serotonin or norepinephrine reuptake inhibitor (SSRI or SNRI) within 4 weeks prior to the start of the trial
* Has a medical or psychiatric condition which compromises the patient's ability to give informed consent or appropriately complete the pain assessments.
* Has an abnormal clinically significant EEG and/or an EEG indicating possible seizure(-like) disorder according to the following abnormalities (with or without clinical significance):

  * spike and wave activity (epileptiform activity)
  * paroxysmal activity
  * abnormal slowing
  * abnormal beta activity
  * asymmetry right-left and anterior-posterior not within normal limits at screening
* Has had alcohol or caffeine in any form during 24 hours before the surgery
* Has abnormal laboratory results at the screening which in the opinion of the

investigator are exclusionary.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Total Pain Relief Score (TOTPAR) | from 0 to 4 hours

SECONDARY OUTCOMES:
Pain Intensity (PI) on a visual analog scale (VAS), PI difference in VAS from Baseline, PI difference on a categorical scale, PI difference on categorical scale from Baseline, Pain Relief (PR) on a categorical scale, PR Intensity Difference (PRID). | at Baseline, 5, 10, 15, 30, 45, 60, and 90 minutes; and 2 through 8 hours or before rescue medication
Time to rescue medication, time to perceptual and meaningful pain relief (stopwatch), time to onset of analgesia, Peak Pain Intensity Difference (PPID), Peak Pain Relief (PPR). | After surgery
Global evaluation of trial medication on a 5-point categorical scale at 8 hours or just prior to rescue medication | at 8 hours or just prior to rescue medication
TOTPAR | over 2, 6, and 8-hour intervals
Summed pain intensity difference (SPID) calculated using PID categorical scale and PID VAS scale, Summed pain relief intensity difference (SPRID), | Over 2, 4, 6, and 8-hour intervals